Date: September 1, 2021

Title: Comparison Effects Of Blue Prescription Program, Home Exercise Program And Supervised Exercise Approaches On Type 2 Diabetic Women.

Identifiers: NCT05479435

## INFORMED CONSENT FORM

Title of the Study: Comparison Effects Of Blue Prescription Program, Home Exercise Program And Supervised Exercise Approaches On Type 2 Diabetic Women.

Purpose of the Study: We aim to investigate the effectiveness of different exercise approaches in individuals with Type 2 Diabetes.

## Participant Information:

Sixty individuals who volunteer to participate in the study will be randomly divided into three groups. If you agree to participate, you will be evaluated by physiotherapist Arzu Abalay. Within the scope of the study, various evaluations including metabolic variables, bioimpedance analysis, skinfold thickness, body mass index, anthropometric measurements, functional capacity, flexibility, physical activity level, quality of life, depression, balance, and satisfaction will be conducted. These evaluations do not pose any risk, and your personal information will be kept confidential. Participation in this study is voluntary, and no fees will be charged. Additionally, no additional payments or medications will be provided.

## **Intervention Procedures:**

Group 1: Participants will be followed up by a physiotherapist once a week for 12 weeks after evaluation and training, and re-evaluated at the end of the 12th week.

Group 2: Participants will receive a video exercise program in the format and method requested by the participant, after group assessment and training, and will be re-evaluated at the end of the 12th week.

Group 3: Participants will exercise with a physiotherapist three days a week for 12 weeks after group assessment and training, and will be re-evaluated at the end of the 12th week.

## Safety Precautions:

If you experience excessive fatigue, shortness of breath, rapid increase in heart rate, or changes in blood sugar during exercise, please inform your physiotherapist. You have the right to withdraw from the study at any time, or your physiotherapist may exclude you.

Contact Information:

Uzm. Fzt. Arzu Abalay

Email: arzuabalay@hotmail.com

Phone: 05075891917 / 02663738170

Position: